CLINICAL TRIAL: NCT00755131
Title: Effects of Cardiac Rehabilitation on High Mobility Group Box-1 Levels After Acute Myocardial Infarction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Carlo Vigorito, Department of Clinical Medicine, Cardiovascular and Immunological Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: UNINA-15775
Record Dates: First submitted 2008-09-17; First posted 2008-09-18 (Estimated); Results first posted 2010-01-25 (Estimated); Last update posted 2010-02-02 (Estimated); Status verified 2009-12

CONDITIONS: Acute Myocardial Infarction
Keywords: Cardiac Rehabilitation; High Mobility Group Box proteins; Inflammatory markers; Cardiopulmonary Functional Capacity; Maximal Oxygen Consumption; Echocardiography; Left Ventricular Ejection Fraction; Left Ventricular Chambers Dilation; Left Ventricular Remodeling; Left Atrium Remodeling; Cardiac Remodeling; Exercise Training
MeSH Terms: conditions — Ventricular Remodeling | interventions — Cardiac Rehabilitation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Training Group (Experimental): Postinfarction patients undergo 6-month exercise-based Cardiac Rehabilitation Program
  Interventions: Other: Exercise-based Cardiac Rehabilitation program
- Control Group (No Intervention): Postinfarction patients NOT undergoing 6-months exercise-based Cardiac Rehabilitation program

INTERVENTIONS:
Other: Exercise-based Cardiac Rehabilitation program — Trained patients attend the exercise training protocol for 6 months on hospital ambulatory-based regimen 3 times/week. Training sessions are supervised under continuous electrocardiography monitoring by a cardiologist, a physiotherapist and a graduate nurse. Each session is preceded by a 5-min warming-up and followed by a 5-min cooling-down. Exercise is performed for 30 min on a bicycle ergometer with the target of 60-70% of the peak oxygen consumption achieved at the initial symptom-limited cardiopulmonary exercise test. Exercise protocol is performed with a gradual increase in exercise workload until the achievement of the predefined target.
  Other Names: Cardiac Rehabilitation
  Arms: Training Group

SUMMARY:
This purpose of this study is to examine the relationship between HMGB-1 and postinfarction predictors of outcome such as cardiopulmonary and echocardiographic parameters before and after a 6-month exercise-based cardiac rehabilitation program.

DETAILED DESCRIPTION:
Exercise-based Cardiac Rehabilitation after acute myocardial infarction (AMI) has beneficial effects on cardiovascular functional capacity, quality of life, risk factors modification, and morbidity and mortality. Mounting evidences suggest that inflammation plays a key role both on initiation and progression of atherosclerosis. Several markers of systemic inflammation appear to be active effectors in the pathophysiology of athero-thrombotic disease leading to the occurrence of AMI.

The high mobility group box 1 (HMGB-1) is a ubiquitous nuclear protein constitutively expressed in quiescent cells, and it has been implicated in several cellular functions, including determination of nucleosomal structure and stability, and binding of transcription factors to DNA sequences. HMGB-1 has been recently recognized as a critical mediator of inflammatory diseases. In fact, the passive release of this protein from necrotic or damaged cells represents an effective stimulus triggering the inflammatory response. Specifically, HMGB-1 binds to the receptor for advanced glycation end products (RAGE) and, in turns, it activates mitogen-activated protein-kinase (MAPK) and nuclear factor-κB (NF-κB).

This intracellular pathway leads to the production of several pro-inflammatory cytokines. Interestingly, increased levels of HMGB-1 have been observed in atherosclerotic lesions, suggesting that HMGB-1 might be involved in the pathophysiology of atherosclerosis.

This study was designed to investigate the relationship between HMGB-1 and strong postinfarction predictors of outcome such as cardiopulmonary and echocardiographic parameters before and after a 6-month exercise-based Cardiac Rehabilitation program.

ELIGIBILITY:
Inclusion Criteria:

* Acute Myocardial Infarction

Exclusion Criteria:

* BMI higher than 30 and lower than 18
* Residual myocardial ischemia
* Severe ventricular arrhythmias
* IIb or III degree atrio-ventricular block
* Valvular disease requiring surgery
* Pericarditis
* Severe renal dysfunction (i.e. creatinine >2.5 mg/dl)
* Severe concomitant non-cardiac disease such as cancer
* Liver dysfunction (alanine aminotransferase/aspartate aminotransferase level >1.5 times the upper normal limit)
* Dementia
* Any systemic disease limiting exercise
* Inability to participate in a prospective study for any logistic reason

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2008-09; Primary Completion 2009-06 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Vigorito, M.D., Study Director — Federico II University
Locations (1):
- University of Naples "Federico II", Naples, Italy

REFERENCES:
- [Background] Giallauria F, Cirillo P, Lucci R, Pacileo M, De Lorenzo A, D'Agostino M, Moschella S, Psaroudaki M, Del Forno D, Orio F, Vitale DF, Chiariello M, Vigorito C. Left ventricular remodelling in patients with moderate systolic dysfunction after myocardial infarction: favourable effects of exercise training and predictive role of N-terminal pro-brain natriuretic peptide. Eur J Cardiovasc Prev Rehabil. 2008 Feb;15(1):113-8. doi: 10.1097/HJR.0b013e3282f00990. PMID 18277196
- [Background] Giallauria F, Galizia G, Lucci R, D'Agostino M, Vitelli A, Maresca L, Orio F, Vigorito C. Favourable effects of exercise-based Cardiac Rehabilitation after acute myocardial infarction on left atrial remodeling. Int J Cardiol. 2009 Aug 21;136(3):300-6. doi: 10.1016/j.ijcard.2008.05.026. Epub 2008 Aug 3. PMID 18676038
- [Background] Giallauria F, De Lorenzo A, Pilerci F, Manakos A, Lucci R, Psaroudaki M, D'Agostino M, Del Forno D, Vigorito C. Reduction of N terminal-pro-brain (B-type) natriuretic peptide levels with exercise-based cardiac rehabilitation in patients with left ventricular dysfunction after myocardial infarction. Eur J Cardiovasc Prev Rehabil. 2006 Aug;13(4):625-32. doi: 10.1097/01.hjr.0000209810.59831.f4. PMID 16874155
- [Background] Giallauria F, De Lorenzo A, Pilerci F, Manakos A, Lucci R, Psaroudaki M, D'Agostino M, Del Forno D, Vigorito C. Long-term effects of cardiac rehabilitation on end-exercise heart rate recovery after myocardial infarction. Eur J Cardiovasc Prev Rehabil. 2006 Aug;13(4):544-50. doi: 10.1097/01.hjr.0000216547.07432.fb. PMID 16874143
- [Background] Giallauria F, Lucci R, Pietrosante M, Gargiulo G, De Lorenzo A, D'Agostino M, Gerundo G, Abete P, Rengo F, Vigorito C. Exercise-based cardiac rehabilitation improves heart rate recovery in elderly patients after acute myocardial infarction. J Gerontol A Biol Sci Med Sci. 2006 Jul;61(7):713-7. doi: 10.1093/gerona/61.7.713. PMID 16870634
- [Background] Cirillo P, Golino P, Calabro P, Cali G, Ragni M, De Rosa S, Cimmino G, Pacileo M, De Palma R, Forte L, Gargiulo A, Corigliano FG, Angri V, Spagnuolo R, Nitsch L, Chiariello M. C-reactive protein induces tissue factor expression and promotes smooth muscle and endothelial cell proliferation. Cardiovasc Res. 2005 Oct 1;68(1):47-55. doi: 10.1016/j.cardiores.2005.05.010. PMID 16023093
- [Background] Cirillo P, Cali G, Golino P, Calabro P, Forte L, De Rosa S, Pacileo M, Ragni M, Scopacasa F, Nitsch L, Chiariello M. Tissue factor binding of activated factor VII triggers smooth muscle cell proliferation via extracellular signal-regulated kinase activation. Circulation. 2004 Jun 15;109(23):2911-6. doi: 10.1161/01.CIR.0000129312.43547.08. Epub 2004 Jun 1. PMID 15173027
- [Background] Libby P, Ridker PM, Maseri A. Inflammation and atherosclerosis. Circulation. 2002 Mar 5;105(9):1135-43. doi: 10.1161/hc0902.104353. PMID 11877368
- [Background] Yamada S, Maruyama I. HMGB1, a novel inflammatory cytokine. Clin Chim Acta. 2007 Jan;375(1-2):36-42. doi: 10.1016/j.cca.2006.07.019. Epub 2006 Jul 25. PMID 16979611
- [Background] Giallauria F, Cirillo P, Lucci R, Pacileo M, D'Agostino M, Maietta P, Vitelli A, Chiariello M, Vigorito C. Autonomic dysfunction is associated with high mobility group box-1 levels in patients after acute myocardial infarction. Atherosclerosis. 2010 Jan;208(1):280-4. doi: 10.1016/j.atherosclerosis.2009.07.025. Epub 2009 Jul 14. PMID 19651408
- [Background] Giallauria F, Cirillo P, Lucci R, Pacileo M, D'agostino M, Maietta P, Vitelli A, Chiariello M, Vigorito C. Effects of exercise-based cardiac rehabilitation on high mobility group box-1 levels after acute myocardial infarction: rationale and design. J Cardiovasc Med (Hagerstown). 2009 Aug;10(8):659-63. doi: 10.2459/JCM.0b013e32832d4979. PMID 19451831
- [Derived] Giallauria F, Cirillo P, D'agostino M, Petrillo G, Vitelli A, Pacileo M, Angri V, Chiariello M, Vigorito C. Effects of exercise training on high-mobility group box-1 levels after acute myocardial infarction. J Card Fail. 2011 Feb;17(2):108-14. doi: 10.1016/j.cardfail.2010.09.001. Epub 2010 Oct 29. PMID 21300299

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was a single-center, randomized, controlled study carried out from October 2008 to January 2009 at the Department of Clinical Medicine, Cardiovascular and Immunological Sciences, University of Naples "Federico II".
Groups:
- Exercise Training Group: Postinfarction patients undergoing 6-month exercise-based Cardiac Rehabilitation Program
- Control Group: Postinfarction patients NOT enrolled in exercise-based Cardiac Rehabilitation program.
Period: Overall Study
Arm/Group | Exercise Training Group | Control Group
Started | 37 | 38
Completed | 37 | 38
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exercise Training Group | Control Group | Total
Number analyzed (Participants) | 37 | 38 | 75
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 28 | 29 | 57
  >=65 years | 9 | 9 | 18
Age Continuous [Mean (Standard Deviation); unit: years] | 60.8 (7.0) | 59.5 (7.7) | 60.4 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 6 | 15
  Male | 28 | 32 | 60
Region of Enrollment [Number; unit: participants]
  Italy | 37 | 38 | 75

OUTCOME MEASURES:

1. Primary Outcome: High Mobility Group Box-1 (HMGB1)Levels at Baseline and 6 Months
Description: High mobility group box-1 (HMGB1) is a ubiquitous nuclear protein, constitutively expressed in quiescent cells, where it is involved in several cellular functions, including determination of nucleosomal structure and stability, and binding of transcription factors to DNA sequences. HMGB1 has been recently recognized as a critical mediator of inflammatory processes: the passive release of this protein from necrotic or damaged cells represents an effective stimulus triggering the inflammatory response.
Time Frame: baseline and 6-month follow-up
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Exercise Training Group | Control Group
Number analyzed (Participants) | 37 | 38
ng/ml
  Baseline | 27.6 (27.8) | 24.5 (18.6)
  6 months | 11.7 (7.0) | 20.5 (15.6)
Statistical Analysis 1: Comparison: Exercise Training Group vs Control Group; Sample size determination was based on a t-test assuming a normal distribution with non-equal variance with the mean and standard deviation for the experimental group (postinfarction patients) of HMGB1 levels equal to 15 ± 7 and 2 ± 1 ng/dl for the control group derived from a previous study, respectively. The required sample size was calculated to be 30 subjects per group to detect on the size of one SD with α value of 0.05 (two-sided) and power (1 - β) of 0.8; Test type: Superiority or Other; p < 0.05, t-test, 2 sided

2. Secondary Outcome: Peak Oxygen Consumption (VO2peak) at Baseline and 6 Months
Description: Oxygen consumption at peak exercise stress testing (VO2peak) was obtained breath-by-breath with use of a computerized metabolic cart. VO2peak was recorded as the mean value of VO2 during the last 20 s of the test and expressed in millilitres per kilogram per minute.
Time Frame: Baseline and 6-month follow-up
Population: intention to treat (ITT) analysis
Measure: Mean (Standard Deviation); unit: ml/kg/min
Arm/Group | Exercise Training Group | Control Group
Number analyzed (Participants) | 37 | 38
ml/kg/min
  baseline | 16.4 (1.5) | 16.7 (2.2)
  6 months | 21.0 (2.4) | 16.3 (1.8)
Statistical Analysis 1: Comparison: Exercise Training Group vs Control Group; Test type: Superiority or Other; p < 0.05, t-test, 2 sided

3. Other Pre Specified Outcome: Heart Rate Recovery at Baseline and 6 Months
Description: The autonomic nervous system (ANS) is the part of the peripheral nervous system that acts as a control system functioning largely below the level of consciousness, and controls visceral functions. It is subdivided into two subsystems: the parasympathetic (vagal) and sympathetic nervous system.
  Sympatho-vagal imbalance is evaluated by post-exercise Heart Rate Recovery (HRR), defined as the fall in heart rate during the first minute after exercise (beats/min). HRR is a marker of vagal tone which is a powerful predictor of all-cause mortality in patients with coronary artery disease.
Time Frame: baseline and 6 month follow-up
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Exercise Training Group | Control Group
Number analyzed (Participants) | 37 | 38
beats/min
  baseline | 13.4 (1.7) | 13.8 (2.7)
  6 months | 19.7 (3.4) | 12.4 (2.5)
Statistical Analysis 1: Comparison: Exercise Training Group vs Control Group; Test type: Superiority or Other; p < 0.05, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | Exercise Training Group | Control Group
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/38
Other Adverse Events (participants affected / at risk) | 0/37 | 0/38

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes